CLINICAL TRIAL: NCT02633293
Title: An Open-Label Extension Study of Inhaled Treprostinil in Subjects With Pulmonary Hypertension Due to Parenchymal Lung Disease
Brief Title: An Open Label Extension Study to Evaluate Inhaled Treprostinil in Adult PH With ILD Including CPFE
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Inhaled treprostinil became commercially available in the US following its approval for PH-ILD
Sponsor: United Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RIN-PH-202
Record Dates: First submitted 2015-12-11; First posted 2015-12-17 (Estimated); Results first posted 2022-12-02 (Actual); Last update posted 2022-12-02 (Actual); Status verified 2022-11

CONDITIONS: Pulmonary Hypertension; Interstitial Lung Disease; Combined Pulmonary Fibrosis and Emphysema
Keywords: Treprostinil; PH; ILD; CPFE; 6 Minute Walk Test
MeSH Terms: conditions — Hypertension, Pulmonary; Lung Diseases, Interstitial; Emphysema | interventions — treprostinil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Inhaled Treprostinil (Experimental): Open-label access
  Interventions: Drug: Inhaled Treprostinil

INTERVENTIONS:
Drug: Inhaled Treprostinil — Inhaled treprostinil up to 15 breaths (90 mcg) four times daily
  Other Names: Tyvaso

SUMMARY:
This is a multicenter, open-label trial to evaluate the safety and efficacy of inhaled treprostinil in subjects with pre-capillary pulmonary hypertension (PH) associated with interstitial lung disease (ILD) including combined pulmonary fibrosis and emphysema (CPFE). The study will include about 266 patients who completed all required assessments in the RIN-PH-201 study at approximately 100 clinical trial centers. The study will continue Your participation in this study is voluntary and will last until you discontinue from the study or the study ends. The study will continue until each subject reaches the Week 108 visit or until inhaled treprostinil become commercially available for patients with PH associated with ILD including CPFE (whichever is sooner).

ELIGIBILITY:
Inclusion Criteria:

1. Subject voluntarily gives informed consent to participate in the study.
2. The subject participated in study RIN-PH-201, remained on study drug, was compliant with RIN-PH-201 study procedures or was enrolled in study RIN-PH-201 at the time that the study was discontinued by the sponsor.
3. Females of reproductive potential must be non-pregnant (as confirmed by a urine pregnancy test at Baseline) and non-lactating, and will:

   * Either abstain from intercourse (when it is in line with their preferred and usual lifestyle), or
   * Use two medically acceptable, highly-effective forms of contraception for the duration of study, and at least 30 days after discontinuing study drug.
4. Males must use a condom for the duration of treatment and for at least 48 hours after discontinuing study drug.

Exclusion Criteria:

1. The subject is pregnant or lactating.
2. The subject was prematurely discontinued from study RIN-PH-201.
3. The subject developed a concurrent illness or condition during the conduct of RIN-PH-201 which, in the opinion of the Investigator, would represent a risk to overall health if they enrolled in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 243 (Actual)
Dates: Start 2016-09-15 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2021-08-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (92):
- United States (91):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - IMC-Diagnostic & Medical Clinic, Mobile, Alabama
  - Arizona Pulmonary Specialists, Ltd., Phoenix, Arizona
  - University of Arizona, Tucson, Arizona
  - Cedars-Sinai Medical Center, Beverly Hills, California
  - University of California, San Francisco-Fresno, Fresno, California
  - University of California San Diego, La Jolla, California
  - VA Long Beach Healthcare System, Long Beach, California
  - University of Southern California, Los Angeles, California
  - Department of Veterans Affairs Greater Los Angeles Healthcare System, Los Angeles, California
  - Pacific Pulmonary Medical Group, Riverside, California
  - University of California Davis Medical Center, Sacramento, California
  - Kaiser Permanente, San Francisco, California
  - University of Colorado Hospital - Cardiac and Vascular Center, Aurora, Colorado
  - National Jewish Health, Denver, Colorado
  - Georgetown University Hospital, Washington D.C., District of Columbia
  - MedStar Heart & Vascular Institute, Washington D.C., District of Columbia
  - Florida Lung, Asthma & Sleep Specialists, P.A., Celebration, Florida
  - St. Francis Sleep, Allergy and Lung Institute, Clearwater, Florida
  - University of Florida Clinical Research Center, Gainesville, Florida
  - University of Florida College of Medicine, Jacksonville, Jacksonville, Florida
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - St. Vincent's Lung, Sleep, and Critical Care Specialists, Jacksonville, Florida
  - University of Miami, Miami, Florida
  - Florida Hospital, Orlando, Florida
  - University of South Florida, Tampa, Florida
  - Cleveland Clinic Florida, Weston, Florida
  - The Emory Clinic, Atlanta, Georgia
  - Piedmont - Georgia Lung Associates, Austell, Georgia
  - Wellstar Medical Group, Marietta, Georgia
  - Northwestern University, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - University of Illinois at Chicago Hospital, Chicago, Illinois
  - University of Chicago Medical Center, Chicago, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Indiana University Hospital, Indianapolis, Indiana
  - Community Heart and Vascular Hospital, Indianapolis, Indiana
  - St. Vincent Medical Group, Inc., Indianapolis, Indiana
  - University of Iowa Hospitals & Clinics, Iowa City, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - University of Louisville Physicians Outpatient Center, Louisville, Kentucky
  - Louisiana State University Health Sciences Center New Orleans, New Orleans, Louisiana
  - Maine Medical Center, South Portland, Maine
  - University of Maryland Medical Center, Baltimore, Maryland
  - Johns Hopkins University, Baltimore, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Spectrum Health Medical Center, Grand Rapids, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - Washington University Hospital, St Louis, Missouri
  - The University of New Mexico, Albuquerque, New Mexico
  - Albany Medical College, Albany, New York
  - New York Methodist Hospital, Brooklyn, New York
  - Northwell Health, New Hyde Park, New York
  - NYU Langone Medical Center, New York, New York
  - The Mount Sinai Hospital, New York, New York
  - Weill Cornell Medical Center, New York, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Pinehurst Medical Clinic, Inc., Pinehurst, North Carolina
  - The Carl and Edyth Lindner Research Center at The Christ Hospital, Cincinnati, Ohio
  - University of Cincinnati Health, Cincinnati, Ohio
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - The Ohio State University Medical Center, Columbus, Ohio
  - Integris Baptist Medical Center, Oklahoma City, Oklahoma
  - Hospital of University of Pennsylvania, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - AnMed Health Pulmonary and Sleep Medicine, Anderson, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Statcare Pulmonary Consultants, Knoxville, Tennessee
  - Baylor University Medical Center at Dallas, Dallas, Texas
  - UT Southwestern Medical Center, Dallas, Texas
  - Texas Tech University Health Sciences Center, El Paso, Texas
  - Houston Methodist, Houston, Texas
  - Michael E. DeBakey VA Medical Center, Houston, Texas
  - The University of Texas Health Science Center at Houston, Houston, Texas
  - The University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - University of Vermont, Vermont Lung Center, Colchester, Vermont
  - Inova Fairfax Hospital, Fairfax, Virginia
  - Sentara Cardiovascular Research Institute, Norfolk, Virginia
  - Pulmonary Associates of Richmond, Richmond, Virginia
  - University of Washington Medical Center, Seattle, Washington
  - University of Wisconsin School of Medicine and Public Health, Madison, Wisconsin
  - Aurora St. Luke's Medical Center, Milwaukee, Wisconsin
  - Medical College of Wisconsin/Froedtert Hospital, Milwaukee, Wisconsin
- Alliance Cardio Pulmonary Research Group, Inc., Guaynabo, Puerto Rico

RESULTS

PARTICIPANT FLOW:
Groups:
- Inhaled Treprostinil: Open-label access
  Inhaled Treprostinil: Inhaled treprostinil (6 mcg/breath) administered four times daily and titrated up to a maximum of 12 breaths four times daily
Period: Overall Study
Arm/Group | Inhaled Treprostinil
Started | 243
Received Inhaled Treprostinil in RIN-PH-202 (Safety Population) | 242
Completed | 70
Not Completed | 173
Not completed — Death | 56
Not completed — Progressive Disease | 12
Not completed — Adverse Event | 29
Not completed — Withdrawal by Subject | 41
Not completed — Protocol Violation | 1
Not completed — Lost to Follow-up | 1
Not completed — Study Terminated by Sponsor | 24
Not completed — Withdrawal by Sponsor Prior to Dose Administration | 1
Not completed — Lung Transplant | 5
Not completed — Lack of Efficacy | 2
Not completed — Principal Investigator Terminated Study Site | 1

BASELINE CHARACTERISTICS:
Population: Safety Population
Arm/Group | Inhaled Treprostinil
Number analyzed (Participants) | 242
Age, Continuous [Median (Full Range); unit: years] | 70.0 [27 to 90]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 116
  Male | 126
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 17
  Not Hispanic or Latino | 224
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3
  Asian | 8
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 53
  White | 178
  More than one race | 0
  Unknown or Not Reported | 0
Time Since Diagnosis [Median (Full Range); unit: years] | 0.51 [0.3 to 13.3]
Current Diagnosis [Count of Participants; unit: Participants]
  Idiopathic interstitial pneumonia | 108
  Chronic hypersensitivity pneumonitis | 13
  Occupational lung disease | 5
  Combined pulmonary fibrosis and emphysema | 59
  Connective tissue disease | 57
6-Minute Walk Distance (6MWD) [Median (Full Range); unit: meters] — Population: Only 229 subjects had a Baseline 6MWD
  meters
    number analyzed (Participants) | 229
    (all) | 270.0 [24 to 549]
N-terminal Pro-brain Natriuretic Peptide (NT-proBNP) [Median (Full Range); unit: pg/mL] — Population: Only 240 subjects had a Baseline NT-proBNP measurement
  pg/mL
    number analyzed (Participants) | 240
    (all) | 465.70 [10.2 to 92,852]
Pulmonary Vascular Resistance [Median (Full Range); unit: Wood units] | 5.100 [3.06 to 18.05]
Mean Pulmonary Artery Pressure [Median (Full Range); unit: mmHg] | 34.5 [25 to 74]
Pulmonary Capillary Wedge Pressure [Median (Full Range); unit: mmHg] | 10.0 [1 to 20]

OUTCOME MEASURES:

1. Primary Outcome: Change in Peak 6-Minute Walk Distance (6MWD) From Baseline
Description: The intent of the 6MWD test is to evaluate exercise capacity associated with carrying out activities of daily living. Change in 6MWD from Baseline correlates with the current clinical standard for assessing patient functional status in the treatment of PH and is considered an objective measure of patient functional status. Subjects will be instructed to walk down a corridor at a comfortable speed as far as they can manage for 6 minutes. Distance <500 meters suggests considerable exercise limitation; Distance 500-800 meters suggests moderate limitation; Distance >800 meters (with no rests) suggests mild or no limitation. Peak exposure 6MWD will occur by conducting 6MWT within 10 to 60 minutes after the most recent dose of study drug dose.
Time Frame: Baseline through Week 124 in RIN-PH-202 (Combined data from parent study RIN-PH-201 [NCT02630316] and this open-label extension study RIN-PH-202)
Population: Values are combined data from the Safety Populations of parent study RIN-PH-201 (n=326; NCT02630316) and this open-label extension study RIN-PH-202 (n=243) as presented in the RIN-PH-202 CSR over the course of 124 weeks (16-week treatment in RIN-PH-201 and up to 108 weeks in RIN-PH-202). The number of subjects analyzed at each week decreased as only those remaining on RIN-PH-202 who had not discontinued early due to the reasons show in the Participant Flow section were evaluated.
Measure: Median (Full Range); unit: meters
Arm/Group | Inhaled Treprostinil
Number analyzed (Participants) | 296
meters
  Week 4 | 1.5 [-197 to 258]
  Week 8: number analyzed (Participants) | 263
  Week 8 | 5.0 [-259 to 196]
  Week 12: number analyzed (Participants) | 246
  Week 12 | 9.5 [-190 to 192]
  Week 16: number analyzed (Participants) | 241
  Week 16 | 10.0 [-269 to 183]
  Week 20: number analyzed (Participants) | 212
  Week 20 | 12.0 [-189 to 169]
  Week 28: number analyzed (Participants) | 189
  Week 28 | 10.0 [-222 to 175]
  Week 40: number analyzed (Participants) | 139
  Week 40 | 3.0 [-261 to 171]
  Week 52: number analyzed (Participants) | 123
  Week 52 | 3.0 [-223 to 194]
  Week 64: number analyzed (Participants) | 109
  Week 64 | -2.0 [-218 to 178]
  Week 76: number analyzed (Participants) | 103
  Week 76 | -2.0 [-209 to 210]
  Week 88: number analyzed (Participants) | 87
  Week 88 | -5.0 [-180 to 185]
  Week 100: number analyzed (Participants) | 63
  Week 100 | -11.0 [-213 to 196]
  Week 112: number analyzed (Participants) | 56
  Week 112 | -24.0 [-183 to 216]
  Week 124: number analyzed (Participants) | 59
  Week 124 | -16.0 [-287 to 190]

2. Secondary Outcome: Change in Plasma Concentration of N-terminal Pro-Brain Natriuretic Peptide (NT-proBNP) From Baseline
Description: The N-terminal pro-BNP (NT-proBNP) serum concentration is a useful biomarker associated with changes in right heart morphology and function. NT-proBNP serum concentration will be assessed to compare the severity of heart failure at Baseline and each visit through Week 124. Blood for NT-proBNP assessment must be drawn prior to conducting the 6-minute walk test (6MWT).
Time Frame: as for outcome 1
Population: RIN-PH-202 CSR over the course of 124 weeks (16-week treatment in RIN-PH-201 and up to 108 weeks in RIN-PH-202). The number of subjects analyzed at each week decreased as only those remaining on RIN-PH-202 who had not discontinued early due to the reasons show in the Participant Flow section were evaluated.
Measure: Median (Full Range); unit: pg/mL
Arm/Group | Inhaled Treprostinil
Number analyzed (Participants) | 285
pg/mL
  Week 8 | -5.10 [-9704.2 to 34,807.3]
  Week 16: number analyzed (Participants) | 250
  Week 16 | -1.30 [-11,433.0 to 87,148.3]
  Week 64: number analyzed (Participants) | 153
  Week 64 | 10.2 [-10,280.0 to 7306.0]
  Week 124: number analyzed (Participants) | 78
  Week 124 | 31.90 [-4500.2 to 26,197.7]

3. Secondary Outcome: Change in Percent Predicted Forced Vital Capacity (FVC) From Baseline
Description: Change in pulmonary function following inhaled treprostinil therapy will be measured by Forced Vital Capacity (FVC), calculated from a Pulmonary Function Test (PFT) performed at Baseline and Weeks 12, 48, and 108.
Time Frame: Baseline and Weeks 12, 48, and 108
Population: Subjects from the Placebo Group in parent study RIN-PH-201
Measure: Median (Full Range); unit: Percent Predicted FVC
Arm/Group | Inhaled Treprostinil
Number analyzed (Participants) | 121
Percent Predicted FVC
  Week 12 | 0.5 [-16 to 23]
  Week 48 | 2.0 [-10 to 21]
  Week 108 | 3.0 [-13 to 13]

ADVERSE EVENTS:
Time Frame: AEs were recorded throughout the course of the study from the time that each subject signed the ICF until all study assessments were completed, through the time that the study was terminated by the Sponsor (following the approval of inhaled treprostinil for use in patients with PH-ILD), up to 108 weeks.
Description: All AEs were followed until resolution (or return to normal or baseline values), until they were judged by the Investigator to no longer be clinically significant, or for at least 30 days if the AE extended beyond the final study visit. All SAEs were followed until resolution, death, or the subject was lost to follow-up, even if they were ongoing more than 30 days after completion of the final study visit.
Arm/Group | Inhaled Treprostinil
All-Cause Mortality (participants affected / at risk) | 56/242
Serious Adverse Events (participants affected / at risk) | 133/242
Other Adverse Events (participants affected / at risk) | 229/242
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Inhaled Treprostinil (N=242)
Anaemia (Blood and lymphatic system disorders) | 2
Iron deficiency anaemia (Blood and lymphatic system disorders) | 2
Lymphadenitis (Blood and lymphatic system disorders) | 1
Immune thrombocytopenia (Blood and lymphatic system disorders) | 1
Right ventricular failure (Cardiac disorders) | 10
Cardiac failure congestive (Cardiac disorders) | 5
Cardiac failure acute (Cardiac disorders) | 3
Cardio-respiratory arrest (Cardiac disorders) | 2
Acute left ventricular failure (Cardiac disorders) | 1
Atrial fibrillation (Cardiac disorders) | 3
Atrial flutter (Cardiac disorders) | 2
Bradycardia (Cardiac disorders) | 1
Cardiac arrest (Cardiac disorders) | 8
Cor pulmonale acute (Cardiac disorders) | 1
Coronary artery disease (Cardiac disorders) | 1
Coronary artery stenosis (Cardiac disorders) | 1
Pulseless electrical activity (Cardiac disorders) | 1
Sinus node dysfunction (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 1
Tachycardia (Cardiac disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 1
Chronic gastritis (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Diverticulum intestinal (Gastrointestinal disorders) | 1
haemorrhagic (Gastrointestinal disorders) | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1
Incarcerated umbilical hernia (Gastrointestinal disorders) | 1
Melaena (Gastrointestinal disorders) | 1
Oesophageal ulcer (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Lower gastrointestinal (Gastrointestinal disorders) | 1
haemorrhage (Gastrointestinal disorders) | 1
Chest pain (General disorders) | 4
Asthenia (General disorders) | 1
Disease progression (General disorders) | 1
Non-cardiac chest pain (General disorders) | 1
Death (General disorders) | 1
Sudden cardiac death (General disorders) | 1
Cholelithiasis (Hepatobiliary disorders) | 1
Acute hepatic failure (Hepatobiliary disorders) | 1
Pneumonia (Infections and infestations) | 21
Sepsis (Infections and infestations) | 7
Arthritis bacterial (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 1
COVID-19 pneumonia (Infections and infestations) | 2
Clostridium difficile infection (Infections and infestations) | 1
Coccidioidomycosis (Infections and infestations) | 1
Fournier's gangrene (Infections and infestations) | 1
Infective exacerbation of (Infections and infestations) | 1
bronchiectasis (Infections and infestations) | 1
Influenza (Infections and infestations) | 3
Metapneumovirus infection (Infections and infestations) | 1
Necrotising fasciitis (Infections and infestations) | 1
Pneumonia bacterial (Infections and infestations) | 1
Pulmonary sepsis (Infections and infestations) | 1
Rhinovirus infection (Infections and infestations) | 1
Septic shock (Infections and infestations) | 3
Staphylococcal bacteraemia (Infections and infestations) | 2
Urinary tract infection (Infections and infestations) | 5
Viral upper respiratory tract (Infections and infestations) | 1
infection (Infections and infestations) | 1
COVID-19 (Infections and infestations) | 1
Clostridium difficile colitis (Infections and infestations) | 1
Osteomyelitis (Infections and infestations) | 1
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1
Pneumonia cytomegaloviral (Infections and infestations) | 1
Pneumonia influenzal (Infections and infestations) | 1
Pneumonia viral (Infections and infestations) | 1
Respiratory syncytial virus (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Urosepsis (Infections and infestations) | 1
Fall (Injury, poisoning and procedural complications) | 2
Subdural haematoma (Injury, poisoning and procedural complications) | 4
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1
Femur fracture (Injury, poisoning and procedural complications) | 1
Hip fracture (Injury, poisoning and procedural complications) | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 1
Liver function test increased (Investigations) | 1
Transaminases increased (Investigations) | 1
Platelet count decreased (Investigations) | 1
Fluid overload (Metabolism and nutrition disorders) | 8
Hyperkalaemia (Metabolism and nutrition disorders) | 2
Hypokalaemia (Metabolism and nutrition disorders) | 2
Hyponatraemia (Metabolism and nutrition disorders) | 3
Dehydration (Metabolism and nutrition disorders) | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1
Hypervolaemia (Metabolism and nutrition disorders) | 2
Malnutrition (Metabolism and nutrition disorders) | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 1
Bone cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Follicular lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Chondrosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Syncope (Nervous system disorders) | 6
Carotid artery stenosis (Nervous system disorders) | 1
Cerebrovascular accident (Nervous system disorders) | 3
Embolic stroke (Nervous system disorders) | 1
Hypoaesthesia (Nervous system disorders) | 1
Ischaemic stroke (Nervous system disorders) | 2
Presyncope (Nervous system disorders) | 1
Thrombotic stroke (Nervous system disorders) | 1
Cerebral haemorrhage (Nervous system disorders) | 1
Encephalopathy (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Seizure (Nervous system disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 9
Nephrolithiasis (Renal and urinary disorders) | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 28
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 13
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 6
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 8
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 3
Combined pulmonary fibrosis and emphysema (Respiratory, thoracic and mediastinal disorders) | 3
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 3
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 4
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 5
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4
Idiopathic interstitial pneumonia (Respiratory, thoracic and mediastinal disorders) | 1
Lung cyst (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 1
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 2
Intertrigo (Skin and subcutaneous tissue disorders) | 1
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 1
Atrial appendage closure (Surgical and medical procedures) | 1
Hypotension (Vascular disorders) | 4
Deep vein thrombosis (Vascular disorders) | 1
Hypertension (Vascular disorders) | 1
Orthostatic hypotension (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Inhaled Treprostinil (N=242)
Cough (Respiratory, thoracic and mediastinal disorders) | 65
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 63
Headache (Nervous system disorders) | 45
Diarrhoea (Gastrointestinal disorders) | 37
Dizziness (Nervous system disorders) | 36
Upper respiratory tract infection (Infections and infestations) | 34
Nausea (Gastrointestinal disorders) | 32
Fatigue (General disorders) | 32
Pneumonia (Infections and infestations) | 30
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 30
Urinary tract infection (Infections and infestations) | 27
Back pain (Musculoskeletal and connective tissue disorders) | 26
Productive cough (Respiratory, thoracic and mediastinal disorders) | 25
Chest pain (General disorders) | 24
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 24
Arthralgia (Musculoskeletal and connective tissue disorders) | 22
Oedema peripheral (General disorders) | 20
Nasopharyngitis (Infections and infestations) | 20
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 19
Sinusitis (Infections and infestations) | 18
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 17
Syncope (Nervous system disorders) | 16
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 16
Bronchitis (Infections and infestations) | 15
Right ventricular failure (Cardiac disorders) | 14
Fluid overload (Metabolism and nutrition disorders) | 14
Pain in extremity (Musculoskeletal and connective tissue disorders) | 14
Acute kidney injury (Renal and urinary disorders) | 14
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 14
Vomiting (Gastrointestinal disorders) | 13
Fall (Injury, poisoning and procedural complications) | 13
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 13
Muscle spasms (Musculoskeletal and connective tissue disorders) | 12
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 12
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institution and/or Principal Investigator agree not to publish or publicly present any results of the Study without the prior written consent of Sponsor, not to be unreasonably withheld or delayed. Institution and/or Principal Investigator further agree to provide Sponsor with drafts of any such publication or presentation for review and approval no less than 30 days prior to submission for publication or the date of public presentation.

DOCUMENTS (2):
  • Study Protocol (2016-08-18): https://cdn.clinicaltrials.gov/large-docs/93/NCT02633293/Prot_000.pdf
  • Statistical Analysis Plan (2019-10-21): https://cdn.clinicaltrials.gov/large-docs/93/NCT02633293/SAP_001.pdf